CLINICAL TRIAL: NCT03353870
Title: Requests for Euthanasia and Assisted Suicide in Establishment of Accommodation for Dependent Old Persons.
Acronym: DESAGE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Principal Investigator, Régis AUBRY, Professor, Centre Hospitalier Universitaire de Besancon
Other Study IDs: Régis Aubry
Record Dates: First submitted 2017-11-13; First posted 2017-11-27 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Qualitative Research; Euthanasia; Assisted Suicide; Aging
MeSH Terms: conditions — Suicide, Assisted

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- qualitative interview: This study has only one arm
  Interventions: Other: qualitative interview

INTERVENTIONS:
Other: qualitative interview — individual qualitative interview

SUMMARY:
The main aim of this project is to analyze and understand the meaning of explicit requests to hasten death (euthanasia and assisted suicide) from older people living in an Establishment of accommodation for dependent old persons.

This involves conducting interviews with patients, carers to whom the request has been expressed and a relative chosen by the patient. This study aims to describe the request over time. This will be done through two series of interviews, one as soon as it is first expressed, then one week later.

ELIGIBILITY:
Inclusion Criteria:

* They live in an establishment of accommodation for dependent old persons
* They have to be ill.
* They have request for euthanasie or assisted suicide
* They are in capacity to meet researchers for interview,
* They aggreed to make an individual interview
* They are covered by the French social security system

Exclusion Criteria:

* They have neurocognitives disorders that can't allow an individual interview
* They did not express themselves a request for euthanasia ou assisted suicide
* They disagreed to participate

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Person living in an establishment of accomation for dépendent old person and requesting an euthanasia.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Qualitative analyse | One year
  Describe, analyze and understand the content, the meaning and factors of evolution of euthanasia or assisted suicide's requests, by crossing the speech of residents, caregivers and family.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Investigation Center, Besançon, Bourgogne-Franche-Comté, France

IPD SHARING:
Plan to Share IPD: No